CLINICAL TRIAL: NCT02519244
Title: Wearable Lower Extremity Exoskeleton to Promote Walking in Persons With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Multiple Sclerosis Society (Other); Texas Woman's University (Other)
Responsible Party: Principal Investigator, Shuo-Hsiu Chang, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HSC-MS-15-0278; PP3394 (Other Grant/Funding Number: National Multiple Sclerosis Society)
Record Dates: First submitted 2015-08-05; First posted 2015-08-10 (Estimated); Results first posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Ambulation; Rehabilitation; Wearable Robotic Devices
MeSH Terms: conditions — Multiple Sclerosis

ARMS (1):
- Robot-assisted rehabilitation (Experimental): Subjects will participate in individualized locomotion training sessions using wearable lower limb exoskeleton, Ekso®. Each training session will last up to 60 minutes, 5 days per week for 3 weeks, for a total of 15 sessions. During the training, subjects will wear a lower extremity exoskeleton robotic walking device. Subjects will participate in individualized treatment sessions which may include: sit to stand, static and dynamic standing balance, weight shifting, walking, turning, and stand to sit.
  Interventions: Device: Ekso® (Wearable lower limb exoskeleton)

INTERVENTIONS:
Device: Ekso® (Wearable lower limb exoskeleton) — The wearable lower limb exoskeleton is a powered, robotic lower limb exoskeleton with actuated hips and knees. A control algorithm has been implemented in this device, which allows for provision of assistance to lower limb segments during movement, dependent on user needs.

SUMMARY:
The purpose of this study is to investigate whether a wearable robotic exoskeleton can help people with multiple sclerosis (MS) to walk again.

DETAILED DESCRIPTION:
Loss of the ability to walk is one of the significant problems in persons with multiple sclerosis (MS). This limitation prevents the person from having an active and meaningful life at home and in the community. Also, more energy is needed to walk, which can cause fatigue and further leads to a non-active life style and poor quality of life. Unfortunately, walking training is often not available for this population because of the severity and progress of the disease; therefore, a new strategy is needed to help people with MS to walk again. A new technology, the wearable robotic exoskeleton, has been developed to help persons with spinal cord injuries stand up and walk. The robotic legs are powered by batteries and controlled by motors. This study will investigate the use of a wearable robotic exoskeleton to help persons with MS to walk. Participants will receive trainings (5 days per week for 3 weeks) to walk with the robotic exoskeleton (EKSO, EKSO Bionics, Richmond, CA). During the training, a physical therapist will teach the participant how to maintain balance, sit to stand, stand to sit, and walk with the wearable robotic exoskeleton. The hypothesis is that persons with MS will be able to use a robotic exoskeleton to walk better and with less energy costs.

ELIGIBILITY:
Subjects will be enrolled if they meet the following inclusion criteria:

* Age 18 years or older
* Ambulatory with assistive devices (Ambulation status will be determined by the EDSS score)
* With an Expanded Disability Status Scale (EDSS) score between 6 and 7.5 inclusive
* Height and weight are between 160 and 188 cm (5'2'' to 6'2''), and less than 100 kg (220 lb), respectively (per exoskeleton manufacturer)
* Able to follow simple 3 step commends
* Able to understand the study procedure and consent form

Subjects will be excluded if they have any of the following exclusion criteria:

* History of severe neurologic injuries other than MS (Spinal Cord Injury, Cerebral Palsy, Amyotrophic Lateral Sclerosis, Traumatic Brain Injury, Cerebral Vascular Accident, etc.)
* Severe comorbidities:

  * active infections
  * heart, lung, or circulatory conditions
  * pressure ulcers
* Documented severe osteoporosis affecting the hip and spine
* Severe spasticity in the lower extremities (Modified Ashworth ≥ 3) or uncontrolled clonus
* Unhealed limb or pelvic fractures
* Skin issues that would prevent wearing the device
* Range of motion restrictions that would prevent subject from achieving a normal, reciprocal gait pattern, or would restrict a subject from completing normal sit to stand or stand to sit transitions.
* Upper extremity strength deficits that limit ability to balance with a front rolling walker or crutches.
* Heterotopic ossification that resists functional range of motion in lower extremities
* Contractures (>15 degrees at the hips or >20 degrees at the knees)
* Psychiatric or cognitive comorbidities resulting in motor planning or impulsivity concerns
* Colostomy
* Have received any physical therapy intervention within 3 months prior to enrolment in the study
* Non-English speaking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-02-06 (Actual); Study Completion 2017-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shuo-Hsiu Chang, PT, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- TIRR Memorial Hermann, Houston, Texas, United States

REFERENCES:
- [Derived] Afzal T, Tseng SC, Lincoln JA, Kern M, Francisco GE, Chang SH. Exoskeleton-assisted Gait Training in Persons With Multiple Sclerosis: A Single-Group Pilot Study. Arch Phys Med Rehabil. 2020 Apr;101(4):599-606. doi: 10.1016/j.apmr.2019.10.192. Epub 2019 Dec 7. PMID 31821798

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 11 were enrolled; however, one person did not initiate the intervention because they were scheduled for knee surgery.
Period: Overall Study
Arm/Group | Robot-assisted Rehabilitation
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Robot-assisted Rehabilitation
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 4
  Asian | 1
  Caucasian | 4
  Hispanic | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10
Weight [Mean (Standard Deviation); unit: kilograms] | 70 (12)
Height [Mean (Standard Deviation); unit: meters] | 1.68 (0.09)
Multiple Sclerosis Type [Count of Participants; unit: Participants]
  Primary Progressive Multiple Sclerosis (PPMS) | 3
  Relapsing-Remitting Multiple Sclerosis (RRMS) | 5
  Secondary Progressive Multiple Sclerosis (SPMS) | 2
Years Since Diagnosis [Mean (Standard Deviation); unit: years] | 15 (7.1)
Kurtzke Expanded Disability Status Scale (EDSS) [Mean (Standard Deviation); unit: units on a scale] — The Kurtzke Expanded Disability Status Scale ranges from 0-10 in increments of 0.5, with higher scores indicating greater severity of disability.
  units on a scale | 6.55 (0.44)

OUTCOME MEASURES:

1. Primary Outcome: Speed in the Timed 25 Feet Walk Test at Self-selected Speed (Without Exoskeleton)
Description: This task will ask the subject to walk for 25 feet at comfortable pace with and without exoskeleton. Subjects will wear their exercise or walking shoes and are allowed to use assistive device such as cane or walker if necessary. The start and finish line of the 25 feet test course will be marked with tape on the floor. Additional 5 feet at the end of start and finish will be used for subject to turn around. A chair will be provided next to the start area so the subject may rest. During the test, the subject will walk at his/her comfortable pace without losing balance. A research team member will walk next to the subject for safety.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: meters per second (m/s)
Arm/Group | Robot-assisted Rehabilitation
Number analyzed (Participants) | 10
meters per second (m/s) | 0.35 (0.18)

2. Primary Outcome: Speed in the Timed 25 Feet Walk Test at Self-selected Speed (Without Exoskeleton)
Description: as for outcome 1
Time Frame: 3 weeks
Population: For two of the subjects not reported, there were technical issues during assessment.
Measure: Mean (Standard Deviation); unit: meters per second (m/s)
Arm/Group | Robot-assisted Rehabilitation
Number analyzed (Participants) | 8
meters per second (m/s) | 0.46 (0.24)

3. Primary Outcome: Speed in the Timed 25 Feet Walk Test at Self-selected Speed (With Exoskeleton)
Description: as for outcome 1
Time Frame: 3 weeks
Population: For two of the subjects not reported, there were technical issues during assessment.
Measure: Mean (Standard Deviation); unit: meters per second (m/s)
Arm/Group | Robot-assisted Rehabilitation
Number analyzed (Participants) | 8
meters per second (m/s) | 0.30 (0.09)

4. Primary Outcome: Speed in the Timed 25 Feet Walk Test at Fast Speed (Without Exoskeleton)
Description: This task will ask the subject to walk for 25 feet at comfortable pace with and without exoskeleton. Subjects will wear their exercise or walking shoes and are allowed to use assistive device such as cane or walker if necessary. The start and finish line of the 25 feet test course will be marked with tape on the floor. Additional 5 feet at the end of start and finish will be used for subject to turn around. A chair will be provided next to the start area so the subject may rest. During the test, the subject will walk at fast speed. A research team member will walk next to the subject for safety.
Time Frame: baseline
Population: One subject did not perform the Timed 25 Feet Walk Test at fast speed because they were only able to walk at the self-selected speed.
Measure: Mean (Standard Deviation); unit: meters per second (m/s)
Arm/Group | Robot-assisted Rehabilitation
Number analyzed (Participants) | 9
meters per second (m/s) | 0.51 (0.24)

5. Primary Outcome: Speed in the Timed 25 Feet Walk Test at Fast Speed (Without Exoskeleton)
Description: as for outcome 4
Time Frame: 3 weeks
Population: One subject did not perform the Timed 25 Feet Walk Test at fast speed because they were only able to walk at the self-selected speed.For one of the subjects not reported, there were technical issues during assessment.
Measure: Mean (Standard Deviation); unit: meters per second (m/s)
Arm/Group | Robot-assisted Rehabilitation
Number analyzed (Participants) | 8
meters per second (m/s) | 0.61 (0.32)

6. Primary Outcome: Speed in the Timed 25 Feet Walk Test at Fast Speed (With Exoskeleton)
Description: as for outcome 4
Time Frame: 3 weeks
Population: For two of the subjects not reported, there were technical issues during assessment.
Measure: Mean (Standard Deviation); unit: meters per second (m/s)
Arm/Group | Robot-assisted Rehabilitation
Number analyzed (Participants) | 8
meters per second (m/s) | 0.33 (0.11)

7. Primary Outcome: Distance Walked During the Six-minute Walk Test (Without Exoskeleton)
Description: Subjects will be asked to walk back and forth in a hallway with or without exoskeleton for 6 minutes. The objective is to cover as much space as possible in 6 minutes. Subjects can slow down or stop to rest if they feel like, but should start walking when they feel they are able. A research team member will walk behind the subject to prevent loss of balance during the test.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Robot-assisted Rehabilitation
Number analyzed (Participants) | 10
meters | 121.15 (64.66)

8. Primary Outcome: Distance Walked During the Six-minute Walk Test (Without Exoskeleton)
Description: as for outcome 7
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Robot-assisted Rehabilitation
Number analyzed (Participants) | 8
meters | 138.90 (66.89)

9. Primary Outcome: Distance Walked During the Six-minute Walk Test (With Exoskeleton)
Description: as for outcome 7
Time Frame: 3 weeks
Population: For two of the subjects not reported, there were technical issues during assessment.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Robot-assisted Rehabilitation
Number analyzed (Participants) | 8
meters | 108.09 (26.26)

10. Primary Outcome: Physical Demands as Assessed by Energy Expenditure (Which is Indicated by VO2-max as Measured by the Cosmed K4b2) During the Timed 25 Feet Walk Test at Self-selected Speed (Without Exoskeleton)
Description: Physical demands during the Timed 25 Feet Walk Test will be indicated by energy expenditure. Energy Expenditure (as indicated by VO2-max) will be measured by the K4 b2 Cosmed as follows: Oxygen cost will be calculated from oxygen consumption as the product of gait speed and body weight. Oxygen consumption will be collected on a breath-by-breath basis measured by a portable metabolic system (K4 b2 Cosmed). Prior to the testing, the system will be calibrated using room air and reference gas mixture. During the testing, the subject will wear a face mask and a heart rate monitor at all times and will be asked to breathe normally.
  VO2-max, also known as maximal oxygen uptake, is the measurement of the maximum amount of oxygen a person can utilize during exercise.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: ml/min/Kg
Arm/Group | Robot-assisted Rehabilitation
Number analyzed (Participants) | 10
ml/min/Kg | 2.83 (1.12)

11. Primary Outcome: Physical Demands as Assessed by Energy Expenditure (Which is Indicated by VO2-max as Measured by the Cosmed K4b2) During the Timed 25 Feet Walk Test at Self-selected Speed (Without Exoskeleton)
Description: as for outcome 10
Time Frame: 3 weeks
Population: For two of the subjects not reported, there were technical issues during assessment.
Measure: Mean (Standard Deviation); unit: ml/min/Kg
Arm/Group | Robot-assisted Rehabilitation
Number analyzed (Participants) | 8
ml/min/Kg | 5.72 (1.06)

12. Primary Outcome: Physical Demands as Assessed by Energy Expenditure (Which is Indicated by VO2-max as Measured by the Cosmed K4b2) During the Timed 25 Feet Walk Test at Self-selected Speed (With Exoskeleton)
Description: as for outcome 10
Time Frame: 3 weeks
Population: For two of the subjects not reported, there were technical issues during assessment.
Measure: Mean (Standard Deviation); unit: ml/min/Kg
Arm/Group | Robot-assisted Rehabilitation
Number analyzed (Participants) | 8
ml/min/Kg | 6.33 (1.32)

13. Primary Outcome: Physical Demands as Assessed by Energy Expenditure (Which is Indicated by VO2-max as Measured by the Cosmed K4b2) During the Timed 25 Feet Walk Test at Fast Speed (Without Exoskeleton)
Description: as for outcome 10
Time Frame: baseline
Population: One subject did not perform the Timed 25 Feet Walk Test at Fast Speed due to fatigue. For another subject, data was not collected for the the Timed 25 Feet Walk Test at Fast Speed due to a technical error.
Measure: Mean (Standard Deviation); unit: ml/min/Kg
Arm/Group | Robot-assisted Rehabilitation
Number analyzed (Participants) | 8
ml/min/Kg | 3.6 (1.31)

14. Primary Outcome: Physical Demands as Assessed by Energy Expenditure (Which is Indicated by VO2-max as Measured by the Cosmed K4b2) During the Timed 25 Feet Walk Test at Fast Speed (Without Exoskeleton)
Description: as for outcome 10
Time Frame: 3 weeks
Population: One subject did not perform the Timed 25 Feet Walk Test at Fast Speed due to fatigue. For another subject, there was a technical error during the assessment.
Measure: Mean (Standard Deviation); unit: ml/min/Kg
Arm/Group | Robot-assisted Rehabilitation
Number analyzed (Participants) | 8
ml/min/Kg | 6.87 (1.44)

15. Primary Outcome: Physical Demands as Assessed by Energy Expenditure (Which is Indicated by VO2-max as Measured by the Cosmed K4b2) During the Timed 25 Feet Walk Test at Fast Speed (With Exoskeleton)
Description: as for outcome 10
Time Frame: 3 weeks
Population: For two of the subjects not reported, there were technical issues during assessment.
Measure: Mean (Standard Deviation); unit: ml/min/Kg
Arm/Group | Robot-assisted Rehabilitation
Number analyzed (Participants) | 8
ml/min/Kg | 7.59 (1.32)

16. Primary Outcome: Physical Demands as Assessed by Energy Expenditure (Which is Indicated by VO2-max as Measured by the Cosmed K4b2) During the Six-Minute Walk Test (Without Exoskeleton)
Description: Physical demands during the Six-Minute Walk Test will be indicated by energy expenditure. Energy Expenditure (as indicated by VO2-max) will be measured by the K4 b2 Cosmed as follows: Oxygen cost will be calculated from oxygen consumption as the product of gait speed and body weight. Oxygen consumption will be collected on a breath-by-breath basis measured by a portable metabolic system (K4 b2 Cosmed). Prior to the testing, the system will be calibrated using room air and reference gas mixture. During the testing, the subject will wear a face mask and a heart rate monitor at all times and will be asked to breathe normally.
  VO2-max, also known as maximal oxygen uptake, is the measurement of the maximum amount of oxygen a person can utilize during exercise.
Time Frame: baseline
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: ml/min/Kg
Arm/Group | Robot-assisted Rehabilitation
Number analyzed (Participants) | 10
ml/min/Kg | 5.76 (1.25)

17. Primary Outcome: Physical Demands as Assessed by Energy Expenditure (Which is Indicated by VO2-max as Measured by the Cosmed K4b2) During the Six-Minute Walk Test (Without Exoskeleton)
Description: as for outcome 16
Time Frame: 3 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: ml/min/Kg
Arm/Group | Robot-assisted Rehabilitation
Number analyzed (Participants) | 8
ml/min/Kg | 10.20 (0.90)

18. Primary Outcome: Physical Demands as Assessed by Energy Expenditure (Which is Indicated by VO2-max as Measured by the Cosmed K4b2) During the Six-Minute Walk Test (With Exoskeleton)
Description: as for outcome 16
Time Frame: 3 weeks
Population: For two of the subjects not reported, there were technical issues during assessment.
Measure: Mean (Standard Deviation); unit: ml/min/Kg
Arm/Group | Robot-assisted Rehabilitation
Number analyzed (Participants) | 8
ml/min/Kg | 7.77 (1.12)

19. Secondary Outcome: Cognitive Demands as Indicated by Reaction Time in Dual Task Paradigm (Without Exoskeleton)
Description: Cognitive demands during the Timed 25 Feet Walk Test at self-selected pace with and without exoskeleton will be determined by reaction time using a dual-task paradigm. We chose a simple reaction time (RT) task, in which the response will be biting on a pressure sensor to make the response pathways as independent as possible from the motor pathways of locomotion. The secondary RT task consists of biting a pressure transducer placed in the mouth in response to an unpredictable sensory (will not cause pain) electrical stimulation applied by an electrode on the back of the neck without changing walking speed and pattern. The stimulation intensity will be adjusted for each individual before data collection. Shorter RT indicates that reduced amount of attentional resources are required.
Time Frame: 3 weeks
Population: For three of the subjects not reported, there were technical issues during assessment.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Robot-assisted Rehabilitation
Number analyzed (Participants) | 7
seconds | 0.51 (0.15)

20. Secondary Outcome: Cognitive Demands as Indicated by Reaction Time in Dual Task Paradigm (With Exoskeleton)
Description: as for outcome 19
Time Frame: 3 weeks
Population: For three of the subjects not reported, there were technical issues during assessment.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Robot-assisted Rehabilitation
Number analyzed (Participants) | 7
seconds | 0.67 (0.43)

21. Secondary Outcome: Amount of Time Taken to Complete the Time Up and Go Test (Without Exoskeleton)
Description: This task will be performed with and without exoskeleton. This task involves subject to stand from the standard chair, walk straight for 3 meters, turn around, walk back to the chair and sit down with shoes and assistive devices if any. A standard chair with arm rests will be place at the start of the testing course. A mark will be placed on the floor at the 3 meter distance.
Time Frame: baseline
Population: One subject was not able to perform the Timed Up and Go test because they required support to sit and stand.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Robot-assisted Rehabilitation
Number analyzed (Participants) | 9
seconds | 33.38 (12.23)

22. Secondary Outcome: Amount of Time Taken to Complete the Time Up and Go Test (Without Exoskeleton)
Description: as for outcome 21
Time Frame: 3 weeks
Population: One subject was not able to perform the Timed Up and Go test because they required support to sit and stand.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Robot-assisted Rehabilitation
Number analyzed (Participants) | 9
seconds | 28.64 (13.74)

23. Secondary Outcome: Quality of Life as Assessed by the Multiple Sclerosis Quality of Life-54 (MSQOL-54) Questionnaire - Physical Health Composite Score
Description: MSQOL-54 physical health composite scores range from 0 to 100, with a higher scale score indicating improved quality of life
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Robot-assisted Rehabilitation
Number analyzed (Participants) | 10
score | 58.3 (12.3)

24. Secondary Outcome: Quality of Life as Assessed by the Multiple Sclerosis Quality of Life-54 (MSQOL-54) Questionnaire - Physical Health Composite Score
Description: as for outcome 23
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Robot-assisted Rehabilitation
Number analyzed (Participants) | 10
score | 57.6 (13.6)

25. Secondary Outcome: Quality of Life as Assessed by the Multiple Sclerosis Quality of Life-54 (MSQOL-54) Questionnaire - Mental Health Composite Score
Description: MSQOL-54 mental health composite scores range from 0 to 100, with a higher scale score indicating improved quality of life
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Robot-assisted Rehabilitation
Number analyzed (Participants) | 10
score | 80.1 (10.7)

26. Secondary Outcome: Quality of Life as Assessed by the Multiple Sclerosis Quality of Life-54 (MSQOL-54) Questionnaire - Mental Health Composite Score
Description: as for outcome 25
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Robot-assisted Rehabilitation
Number analyzed (Participants) | 10
score | 78.8 (13.2)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Robot-assisted Rehabilitation
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
Single arm design; the size range of the exoskeleton limited the inclusion of subjects despite meeting all other inclusion criteria.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-27): https://cdn.clinicaltrials.gov/large-docs/44/NCT02519244/Prot_SAP_000.pdf